CLINICAL TRIAL: NCT03903185
Title: Pharmacokinetics of Ledipasvir/Sofosbuvir in Hepatitis C Virus-Infected Children With Hematological Malignancy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Manal Hamdy El-Sayed, Professor of Pediatrics and Director of the Clinical Research Center, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL 3062
Record Dates: First submitted 2019-04-03; First posted 2019-04-04 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Hepatitis C, Chronic; Hematologic Malignancy
Keywords: Hepatitis C virus; Pharmacokinetic Modeling; Pharmacokinetics; Pediatrics; Leukemia; Ledipasvir; Sofosbuvir; Antiviral Drugs
MeSH Terms: conditions — Hepatitis C, Chronic; Hematologic Neoplasms; Hepatitis C; Leukemia | interventions — ledipasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HCV-infected patients with hematological malignancy (Active Comparator): HCV-infected patients with hematological malignancy on maintenance chemotherapy
  Interventions: Drug: Ledipasvir / Sofosbuvir Oral Product
- Control HCV-infected patients (Active Comparator): Control HCV-infected patients without haematological malignancy or co-morbidities.
  Interventions: Drug: Ledipasvir / Sofosbuvir Oral Product

INTERVENTIONS:
Drug: Ledipasvir / Sofosbuvir Oral Product — 45 mg of ledipasvir and 200 mg of sofosbuvir orally, once daily with food
  Other Names: LDV\SOF

SUMMARY:
This is a prospective, controlled, open-label, pharmacokinetic study. This study aims at studying the PK of ledipasvir, sofosbuvir, and GS-331007 metabolite in HCV infected children with hematological malignancy.

In this study, patients in both treatment groups will receive 12 weeks of treatment with a ﬁxed-dose combination tablet containing 45 mg of ledipasvir and 200 mg of sofosbuvir (LDV/SOF) orally, once daily with food.

DETAILED DESCRIPTION:
In this study, patients in both treatment groups will receive 12 weeks of treatment with a ﬁxed-dose combination tablet containing 45 mg of ledipasvir and 200 mg of sofosbuvir (LDV/SOF) orally, once daily with food, as prescribed by the attending physician.

Twelve eligible HCV-infected patients with hematological malignancy and 12 matching HCV control patients without haematological malignancy or co-morbidities will be enrolled in the study.

At baseline, careful history of the recruited patients including demographic characteristics (age, height, weight, and gender), comorbidities, medication history, familial history, social history, blood transfusion history, time on maintenance chemotherapy, and baseline laboratory tests will be documented. The baseline laboratory tests will include renal function tests (serum creatinine), liver function tests (bilirubin, albumin, AST, and ALT), international normalized ratio (INR), alpha fetoprotein (AFP), complete blood count (CBC), degree of liver fibrosis by Fibroscan, and viral load by PCR.

Followup will be done for all participants at baseline, after 12 weeks of treatment, and after 12 weeks from the end of treatment. A Forth visit will be done after 10 days of treatment for the evaluation of the steady state PK parameters of LDV\SOF in those patients.

ELIGIBILITY:
Inclusion Criteria:

* Children (6 to < 12 years of age and/or weighing 17.5 to < 35 Kg).
* Chronic HCV genotype 4 infection for at least 6 months without cirrhosis (confirmed by Fibroscan).
* Naïve patients to previous anti-HCV treatment.
* Diagnosed with hematological malignancy and on maintenance chemotherapy.

Exclusion Criteria:

* Known hypersensitivity to any of the study medications.
* Ongoing treatment with any interacting medications like carbamazepine, fosphenytoin, phenytoin, oxcarbazepine, phenobarbital, and rifampin.
* History of any comorbid illness that may interfere with the pharmacokinetics of the study drugs or prohibit the compliance with the study protocol such as;

  1. Decompensated liver disease as shown by the presence of ascites, encephalopathy, or a history of variceal hemorrhage.
  2. The ongoing treatment of other types of cancer or blood disorders.
  3. Co-infection with human immunodeficiency virus (HIV), or hepatitis B virus.
  4. Renal dysfunction.
  5. Active infection that is currently producing symptoms.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Measurement of the pharmacokinetics of LDV\SOF | Blood samples will be collected after 10 days of treatment
  After 10 days of treatment, the steady state for LDV/SOF will be reached. Serial blood samples (2 mL/sample) will be collected at this time for the determination of LDV/SOF and GS-331007 concentrations from patients using an eight-point plasma schedule.
  Blood sampling schedule will be as follows (Predose, 0.5,1, 2, 3, 4, 8, and 12h post dose; with predose also serving as t = 24).
  Any deviations from nominal sampling times will be accurately recorded.

SECONDARY OUTCOMES:
Measurement of the number of participants with sustained virological response (SVR12), 12 weeks after discontinuation of therapy with ledipasvir-sofosbuvir (LDV-SOF). | 12 weeks after discontinuation of therapy with ledipasvir-sofosbuvir (LDV\SOF)
  Number of Participants with sustained virological response at 12 Weeks after end of study drug treatment (SVR12) will be recorded.
  Participant will be considered to have achieved SVR12 if HCV RNA is less than the lower limit of quantification of <15 IU/ml) at 12 weeks after the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Manal H Elsayed, MD, Principal Investigator — Ain Shams University
Locations (2):
- Egypt (2):
  - Faculty of Medicine Ain Shams Research Institute- Clinical Research Center (MASRI-CRC), Cairo, Cairo Governorate
  - Pediatric Hematology Oncology and BMT Department, Faculty of Medicine, Ain Shams University, Cairo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] AbdelMagid AM, Abbassi MM, Ebeid FS, El-Sayed MH, Farid SF. Population Pharmacokinetics of Ledipasvir/Sofosbuvir in Pediatric Patients: Impact of Acute Lymphoblastic Leukemia. Clin Ther. 2025 Feb;47(2):e5-e15. doi: 10.1016/j.clinthera.2024.11.022. Epub 2024 Dec 19. PMID 39706761
- [Derived] AbdelMagid AM, Abbassi MM, Ebeid FS, Farid SF, El-Sayed MH. Ledipasvir/Sofosbuvir in Hepatitis C Virus-Infected Children With Hematological Malignancies: A Pharmacokinetic Study. Clin Ther. 2024 Jan;46(1):e12-e22. doi: 10.1016/j.clinthera.2023.10.007. Epub 2023 Nov 3. PMID 37925363